CLINICAL TRIAL: NCT04951167
Title: EFFECT OF DIFFERENT NOREPINPHRINE APPLICATION METHODS IN CAESARIANES ON HYPOTENSION AFTER SPINAL ANESTHESIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Nurşen Seyhun, M.D., Inonu University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-120
Record Dates: First submitted 2021-07-01; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: HYPOTENSION AFTER SPINAL ANESTHESIA,IN PREGNANCY
Keywords: NOREPINPHRINE; SPINAL ANESTHESIA; HYPOTENSION; pregnancy
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Pregnant women will be randomly divided into 4 groups using the closed envelope method. The person who prepares the study drugs and follows the study will be different and unaware of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PB: prophylactic bolus (Active Comparator): an IV bolus of 4 mcg Norepinephrine will be administered immediately after spinal anesthesia, and then SF infusion will be started at 1 ml/min.
  Interventions: Drug: Norepinephrine
- PI:prophylactic infusion (Active Comparator): 1ml of saline is administered immediately after spinal anesthesia, and then infusion will be started with the study drug at 1 ml/min.(4mcg/min)
  Interventions: Drug: Norepinephrine
- TB:therapeutic bolus (Active Comparator): immediately after spinal anesthesia, 1 ml of saline, followed by 1 ml/min infusion of SF, and when the blood pressure decreases by 20%, 1 ml of working solution and then 1 ml/min of saline infusion will be started.
  Interventions: Drug: Norepinephrine
- TBI:therapeutic bolus-infusion (Active Comparator): 1 ml of study drug and 1 ml/min of study drug infusion will be started immediately after spinal anesthesia, after 1 ml of saline followed by 1 ml/min of SF infusion when blood pressure decreases by 20% of the entry
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — in the form of infusion
  Arms: PB: prophylactic bolus; TB:therapeutic bolus; TBI:therapeutic bolus-infusion
Drug: Norepinephrine — in the form of bolus
  Arms: PI:prophylactic infusion; TBI:therapeutic bolus-infusion

SUMMARY:
There are previous studies in which norepinephrine was administered only as a prophylactic or only infusion to prevent hypotension after spinal anesthesia in cesarean sections. However, there are not enough studies reporting which of these application methods are more effective. Therefore, in our study, cesarean section under spinal anesthesia was planned; We aimed to investigate the effectiveness of norepinephrine differential administration methods on preventing maternal hypotension.

DETAILED DESCRIPTION:
EFFECT OF DIFFERENT NOREPINPHRINE APPLICATION METHODS IN CAESARIANES ON HYPOTENSION AFTER SPINAL ANESTHESIA INTRODUCTION Spinal anesthesia in cesarean sections is a frequently used anesthesia technique today. The most common complication associated with spinal anesthesia is hypotension. Systemic vascular resistance and cardiac output decrease due to sympathetic blockade, and when this is accompanied by bradycardia and contractility, hypotension develops(1,2,3).

Maternal hypotension is a condition that can cause negative consequences such as nausea, vomiting, and dizziness in pregnant women who undergo spinal anesthesia. In addition, it increases the likelihood of fetal acidosis, hypoxia, and neonatal neurological damage. Therefore, it is necessary to treat maternal hypotension effectively. In the current treatment of maternal hypotension, intravenous fluid administration, treatments such as ephedrine, phenylephrine, and norepinephrine are used (4,5,7). Among these drugs, ephedrine is the first preferred vasopressor (4). For this reason, its efficacy and safety, and the use of different doses have been extensively studied (5,7). Ephedrine is a vasopressor with both direct and indirect effects in the treatment of hypotension due to neuraxial block in obstetrics with its alpha and beta agonist effects. The most important disadvantage of ephedrine is that it has a slow onset and weak effect, difficulty in titration, development of tachyphylaxis, causing maternal tachy-arrhythmias and fetal acidosis (9). Ephedrine easily crosses the placenta and causes fetal tachycardia, an increase in noradrenaline concentration in the umbilical artery (UA), and a decrease in pH and base excess (BE). An increase in fetal metabolic rate, an increase in fetal O2 consumption and CO2 production, and an increase in lactate level are observed through beta-adrenergic stimulation (9). Phenylephrine, on the other hand, is a pure alpha-agonist agent that is more potent (phenylephrine/ephedrine: 80:1), easy to titrate, effectively treats hypotension and nausea-vomiting, has minimal placental transfer, and does not cause fetal acidosis and changes (10-11). However, the disadvantage of phenylephrine is that it decreases maternal heart rate and cardiac output (12). Another vasopressor drug used in the treatment of hypotension in recent years is norepinephrine. Norepinephrine is both an α-receptor agonist and a weak β-receptor agonist (7,8). Theoretically, it lowers heart rate and cardiac output less.

There are previous studies in which norepinephrine was administered only as a prophylactic or only infusion to prevent hypotension after spinal anesthesia in cesarean sections. However, there are not enough studies reporting which of these application methods are more effective. Therefore, in our study, cesarean section under spinal anesthesia was planned; We aimed to investigate the effectiveness of norepinephrine differential administration methods on preventing maternal hypotension.

WORKING PROTOCOL After the approval of the faculty ethics committee, the written and verbal consent of the patients will be obtained, and a double-blind randomized study will be initiated.

Pregnant women over the age of 18, with ASA (American Society of Anesthesiologists physical status) ≤ III, body weight 50-100 kg and height 150-180 cm, with a single pregnancy planned for cesarean section under elective conditions under spinal anesthesia, will be included in the study.

Pregnant women with allergy or hypersensitivity to norepinephrine, pre-existing hypertension or pregnancy-induced hypertension, cardiovascular or cerebrovascular disease, renal failure, history of thrombosis in the mesenteric or peripheral vessels, history of diabetes with known fetal anomalies, users of monoaminooxidase inhibitors, tricyclic antidepressants and those who refused to study were excluded.

Pregnant women will be randomly divided into 4 groups using the closed envelope method. The person who prepares the study drugs and follows the study will be different and unaware of the study. Following standard aspiration prophylaxis and monitoring, peripheral vascular access will be established with an 18-G catheter and 1 ml/kg/hour Ringer Lactate solution will be started. Basal systolic blood pressure will be determined by measuring heart rate values every 2 minutes and averaging the 3 values.

Spinal anesthesia will be provided in the sitting position with a 25-gauge Quinke spinal needle through the L3-L4 or L4-L5 spacing with 2-2.2 ml of hyperbaric bupivacaine and 15 mcg of fentanyl. Immediately after spinal anesthesia, the pregnant woman will be placed in the supine position, with a pillow placed under the right hip (30 tilts to the left) and rapid coloading with 10 ml/kg Ringer Lactate at a maximum of 1 L with the help of a pump. Afterwards, the mai rate will be reduced to 1 ml/kg/hour again. For the study, norepinephrine will be prepared at 4 mcg/ml.

In Group PB, an IV bolus of 4 mcg will be administered immediately after spinal anesthesia, and then SF infusion will be started at 1 ml/min.

In Group PI, 1ml of saline is administered immediately after spinal anesthesia, and then infusion will be started with the study drugat 1 ml/min.(4mcg/min) In Group TB, immediately after spinal anesthesia, 1 ml of saline, followed by 1 ml/min infusion of SF, and when the blood pressure decreases by 20%, 1 ml of working solution and then 1 ml/min of saline infusion will be started.

In Group TBI, 1 ml of study drug and 1 ml/min of study drug infusion will be started immediately after spinal anesthesia, after 1 ml of saline followed by 1 ml/min of SF infusion when blood pressure decreases by 20% of the entry. Heart rate and blood pressure and pulse oximetry will be recorded every 2 minutes from intrathecal drug administration until delivery. When systolic blood pressure drops more than 20% compared to baseline, it will be considered as hypotension and an additional 4 mcg (1 ml) norepinephrine will be administered in all groups, and if it continues in the next measurement, a second dose of 4 mcg norepinephrine will be administered. Hypotension that does not improve despite two measurements will be treated with an IV bolus of 10 mg of ephedrine. According to entry, 40% or more will be considered severe hypotension and treated with 15 mg of ephedrine. If the heart rate drops to 50 beats/minute, bradycardia will be considered and treated with 0.5 mg of atropine. Hypertension will be considered as a 20% increase in systolic blood pressure from baseline and treated with a 0.1 mg bolus of nitroglycerin iv. The study protocol will be terminated after the delivery of the fetus, but anesthetist bolus norepinephrine administration will be continued for the treatment of hypotension. The number of episodes of hypotension and hypertension, bradycardia, nausea, vomiting, tremor, sensory block level, Apgar score, umbilical artery and vein values, time from intrathecal injection to delivery, uterine incision delivery times will be recorded.

RESOURCES Morgan GE, Mikhail MS, Murray MJ, Larson CP: Clinical Anesthesiology (LANGE), Güneş Bookstore, Third Edition, Ankara, 2004.P:260-269.

2. Kayhan Z: Clinical Anesthesia. Logos Yay.Tic.A.Ş., Second Edition, Istanbul: 1997. P:482-489.

3. Edirne S, Özyalçın SN, Raj PP, Heavner J, Aldemir T, Yücel A: Regional Anesthesia. Nobel Medicine Bookstores, Istanbul 2005. P:159-184.

4. Kinsella S, Carvalho B, Dyer R, et al. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia 2018;73:71-92.

5. Lee A, Ngan Kee WD, Gin T. A quantitative, systematic review of randomized controlled trials of ephedrine versus phenylephrine for the management of hypotension during spinal anesthesia for cesarean delivery. Anesth Analg 2002;94:920-6.

6. Habib AS. A review of the impact of phenylephrine administration on maternal hemodynamics and maternal and neonatal outcomes in women undergoing cesarean delivery under spinal anesthesia. Anesth Analg 2012;114:377-90.

7. Chen D, Qi X, Huang X, et al. Efficacy and safety of different norepinephrine regimens for prevention of spinal hypotension in cesarean section: a randomized trial. Biomed Res Int 2018;2018:2708175.

8. Onwochei DN, Ngan Kee WD, Fung L, et al. Norepinephrine intermittent intravenous boluses to prevent hypotension during spinal anesthesia for cesarean delivery: a sequential allocation dose-finding study. Anesth Analg 2017;125:212-8.

9. Ngan Kee WD, Khaw KS, Tan PE, Ng FF, Karmakar MK. Placental transfer and fetal metabolic effects of phenylephrine and ephedrine during spinal anesthesia for cesarean delivery. Anesthesiology 2009;111:506-12.

10. Ngan Kee WD, Khaw KS, Tan PE, Ng FF, Karmakar MK. Placental transfer and fetal metabolic effects of phenylephrine and ephedrine during spinal anesthesia for cesarean delivery. Anesthesiology 2009;111:506-12.

11. Saravanan S, Kocarev M, Wilson RC, Watkins E, Columb MO, Lyons G. Equivalent dose of ephedrine and phenylephrine in the prevention of post-spinal hypotension in Caesarean section. Br J Anaesth 2006;96:95-9.

12. Cooper D.W. Caesarean delivery vasopressor management. Curr Opin Anaesthesiol 2012; 25:300-8.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women over the age of 18, with ASA (American Society of Anesthesiologists physical status) ≤ III, body weight 50-100 kg and height 150-180 cm, with a single pregnancy planned for cesarean section under elective conditions under spinal anesthesia, will be included in the study.

Exclusion Criteria:

Pregnant women with allergy or hypersensitivity to norepinephrine, pre-existing hypertension or pregnancy-induced hypertension, cardiovascular or cerebrovascular disease, renal failure, history of thrombosis in the mesenteric or peripheral vessels, history of diabetes with known fetal anomalies, users of monoaminooxidase inhibitors, tricyclic antidepressants and those who refused to study were excluded.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
systolic blood pressure | every 2 mins from intrathecal drug administration until delivery
  When systolic blood pressure drops more than 20% compared to baseline, it will be considered as hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Nurcin Gulhas, Prof, Principal Investigator — Inonu Universitesi
Locations (1):
- Inonu Universitesi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Background] Lee A, Ngan Kee WD, Gin T. A quantitative, systematic review of randomized controlled trials of ephedrine versus phenylephrine for the management of hypotension during spinal anesthesia for cesarean delivery. Anesth Analg. 2002 Apr;94(4):920-6, table of contents. doi: 10.1097/00000539-200204000-00028. PMID 11916798
- [Background] Habib AS. A review of the impact of phenylephrine administration on maternal hemodynamics and maternal and neonatal outcomes in women undergoing cesarean delivery under spinal anesthesia. Anesth Analg. 2012 Feb;114(2):377-90. doi: 10.1213/ANE.0b013e3182373a3e. Epub 2011 Nov 21. PMID 22104076
- [Background] Chen D, Qi X, Huang X, Xu Y, Qiu F, Yan Y, Li Y. Efficacy and Safety of Different Norepinephrine Regimens for Prevention of Spinal Hypotension in Cesarean Section: A Randomized Trial. Biomed Res Int. 2018 May 23;2018:2708175. doi: 10.1155/2018/2708175. eCollection 2018. PMID 29951531
- [Background] Onwochei DN, Ngan Kee WD, Fung L, Downey K, Ye XY, Carvalho JCA. Norepinephrine Intermittent Intravenous Boluses to Prevent Hypotension During Spinal Anesthesia for Cesarean Delivery: A Sequential Allocation Dose-Finding Study. Anesth Analg. 2017 Jul;125(1):212-218. doi: 10.1213/ANE.0000000000001846. PMID 28248702
- [Background] Ngan Kee WD, Khaw KS, Tan PE, Ng FF, Karmakar MK. Placental transfer and fetal metabolic effects of phenylephrine and ephedrine during spinal anesthesia for cesarean delivery. Anesthesiology. 2009 Sep;111(3):506-12. doi: 10.1097/ALN.0b013e3181b160a3. PMID 19672175
- [Background] Saravanan S, Kocarev M, Wilson RC, Watkins E, Columb MO, Lyons G. Equivalent dose of ephedrine and phenylephrine in the prevention of post-spinal hypotension in Caesarean section. Br J Anaesth. 2006 Jan;96(1):95-9. doi: 10.1093/bja/aei265. Epub 2005 Nov 25. PMID 16311286
- [Background] Cooper DW. Caesarean delivery vasopressor management. Curr Opin Anaesthesiol. 2012 Jun;25(3):300-8. doi: 10.1097/ACO.0b013e3283530d62. PMID 22473212